CLINICAL TRIAL: NCT04848233
Title: Development of Methodology for Use of Continuous Blood Glucose Measurements When Evaluating Meal Effects on Glucose Regulation - a Pilot Trial
Brief Title: Using CGM for Evaluating Effects of Food on Glucose Regulation in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DoubleGood AB (Industry)
Collaborators: starScience GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DG2101_CGM
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Glycemic Control; Diet, Food and Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drink intervention (Other): Placebo and two drinks containing a blend of five amino acids and chromium picolinate, are included with every main meal and served in a standardized, non-randomised order.
  Interventions: Dietary Supplement: Drinks containing 5AA+CrPic and Placebo

INTERVENTIONS:
Dietary Supplement: Drinks containing 5AA+CrPic and Placebo — Same diet will be repeated for 3 days in a row and the beverage switched every day. 3 periods of 3 days are included in the study.

SUMMARY:
The specific goal of this pilot study is to evaluate if it is possible to detect a statistical difference in postprandial glycemia after meals served with and without a drink previously shown to reduce postprandial glycemia by about 25%. A third drink, with a new recipe, is also included for comparisons. Six participants will carry continuous blood glucose monitors for 10 days and follow a specific meal schedule. The data from this study will form the basis for forming hypothesis of future studies as well as make appropriate calculations of statistical power.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-29.9 kg/m^2
* HOMA-IR < 2.5
* Fasting glucose < 6.1 mmol/L
* Stable weight since 3 months
* Access to iPhone with Bluetooth 4.0 and iOS 13 or later

Exclusion Criteria:

* Diabetes
* Pharmacological treatment known to interfer with metabolism
* Antibiotics treatment the latest 3 months
* Vegetarian/Vegan diet
* Use of tobacco
* Pregnancy or breast-feeding

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose response | From start of meal (0 min) to 120 min postprandially
  Incremental area under the blood glucose curve after each meal

SECONDARY OUTCOMES:
Glycemic variability | 24 hour cycles
  Variation in blood glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Elin Ostman, PhD, Principal Investigator — Aventure AB
Locations (1):
- Aventure AB, Lund, Sweden

REFERENCES:
- [Result] Samigullin A, Humpert PM, Ostman E. Continuous glucose monitoring as a close to real life alternative to meal studies - a pilot study with a functional drink containing amino acids and chromium. Front Med Technol. 2022 Aug 18;4:931837. doi: 10.3389/fmedt.2022.931837. eCollection 2022. PMID 36062264